CLINICAL TRIAL: NCT03543540
Title: A Phase 1 Study of Nexvax2 Administered Subcutaneously After a Screening Gluten Food Challenge That Compares Relative Bioavailability With Intradermal Administration in Non-homozygous HLA-DQ2.5+ Adults With Celiac Disease
Brief Title: Bioequivalence Study of Nexvax2 in Subjects With Celiac Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmusanT, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nexvax2-1005
Record Dates: First submitted 2018-04-26; First posted 2018-06-01 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Celiac Disease; Intestinal Disease; Malabsorption Syndromes; Gastrointestinal Disease; Digestive System Diseases; Metabolic Disease; Coeliac Disease; Gluten Sensitivity
MeSH Terms: conditions — Celiac Disease; Intestinal Diseases; Malabsorption Syndromes; Gastrointestinal Diseases; Digestive System Diseases; Metabolic Diseases | interventions — Nexvax2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Nexvax2 (Arm A) (Experimental)
  Interventions: Biological: Nexvax2
- Nexvax2 (Arm B) (Experimental)
  Interventions: Biological: Nexvax2
- Nexvax2 Placebo (Arm C) (Placebo Comparator)
  Interventions: Biological: Placebo
- Nexvax2 Placebo (Arm D) (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nexvax2 — Nexvax2 injections: 14 in total at twice weekly intervals
  Arms: Nexvax2 (Arm A); Nexvax2 (Arm B)
Biological: Placebo — Placebo injections: 14 in total at twice weekly intervals
  Arms: Nexvax2 Placebo (Arm C); Nexvax2 Placebo (Arm D)

SUMMARY:
A randomized, double-blind, placebo-controlled clinical study in non-homozygous human leukocyte antigen (HLA)-DQ.2.5+ adults with celiac disease (CeD).

DETAILED DESCRIPTION:
A Phase 1, randomized,double-blind, placebo-controlled clinical study of Nexvax2, in adult subjects with confirmed CeD who, have been following a gluten free diet for at least 12 consecutive months prior to screening. The study will evaluate the safety and tolerability of Nexvax2 administered subcutaneously and will compare the bioavailability of subcutaneous versus intradermal administration. The study plan consists of 3 periods: a screening period of 3 to 5 weeks, a 46-day treatment period, and a 30-day post-treatment observational follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 70 years of age (inclusive)
* History of medically diagnosed Celiac Disease (CeD) that included duodenal biopsy.
* Maintenance of gluten free diet (GFD) for at least 12 consecutive months prior to screening.
* Willingness to consume a moderate amount of gluten on one occasion during screening.
* Able to read and understand English.

Exclusion Criteria:

* History of inflammatory bowel disease and/or microscopic colitis.
* Any medical condition or lab abnormality that in the opinion of the investigator may interfere with study conduct or would impact the immune response (other than CeD), confound interpretation of study results, or pose an increased risk to the subject.
* Use of immunomodulatory or immune-suppressing medical treatment during the 6 months prior to screening
* Use of oral or parenteral immunomodulatory corticosteroids, within the 6 weeks prior to screening. Topical or inhaled corticosteroids are acceptable.
* Receipt of any investigational drug or participation in another clinical study within 6 months prior to screening.
* Females who are lactating or pregnant
* Receipt of any vaccine within 1 week prior to planned first day of the treatment period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Safety of Nexvax 2 administered subcutaneously (SQ) | Treatment Period: 7 weeks
  Treatment emergent adverse events (TEAEs) will be summarized by treatment group and treatment arm, severity (grades as defined in CTCAE, Version 4.03), relationship to IP, and phase of treatment and presented as the number and percentage of patients reporting an event(s) as well as the number of events reported.
Evaluate bioavailability of the constituents of Nexvax2 after SQ versus intradermal (ID) administration | Treatment Period: 7 weeks
  Blood draws for plasma concentration

SECONDARY OUTCOMES:
Evaluate the pharmacodynamics (PD) of the maintenance dose levels of Nexvax2 administered SQ and ID | Treatment Period: 7 weeks
  Blood draw collected for cytokines
Evaluate area under the plasma concentration-time curve for the constituents of Nexvax2 in SQ versus ID maintenance doses. | Treatment Period: 7 weeks
  Blood draw collected for Pharmacokinetic (PK) sample
Compare elimination half life properties for the constituents of Nexvax2 in SQ versus ID maintenance doses. | Treatment Period: 7 weeks
  Blood draw collected for PK
Compare time to maximal plasma concentration for the constituents of Nexvax2 in SQ versus ID maintenance doses. | Treatment Period: 7 weeks
  Blood draw collected for PK

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anderson, PhD, FRACP, Study Chair — ImmusanT, Inc.
Locations (3):
- Australia (3):
  - Qpharm Pty Ltd, Herston, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: ImmusanT — http://www.immusant.com/